CLINICAL TRIAL: NCT05782634
Title: Insertion of Immediate Cortical Satellite Implants With Immediate Loading in the Maxillary Esthetic Zone, a Case Series Study
Brief Title: Insertion of Immediate Cortical Satellite Implants With Immediate Loading
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Essam Mohamed Mahmoud, master candidate, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: essam95
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Immediate Loading , Satellite Implant , Immediate Implant
Keywords: immediate loading , satellite implant , immediate implant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subjected to immediate cortical satellite implants with immediate loading (Experimental): All patients involved in this study will be subjected to immediate cortical satellite implants with immediate loading
  Interventions: Device: immediate satellite implant with immediate loading

INTERVENTIONS:
Device: immediate satellite implant with immediate loading — Infiltration anesthesia will be administered using mepivacaine HCl (2%) with levonordefrin 1:20 000 . Injection to control pain and bleeding for hemostasis.
  Dental extraction will be done with minimal force to avoid trauma to the bone. Flab will be released, different drilling sizes will be used to attain the final drill size of the planed implant height and width according to Cone Beam CT. Implants were screwed directly into the osteotomy site, a satellite implant device is attached to the implant's abutment placed on the buccal and palatal plates of bone and retention between the abutment and microplate will help in neglecting the lateral destructive forces . sutures will be done . Impression will be taken for immediate loading with the final crown. Cone beam will be done.

SUMMARY:
Statement of the problem:

Based on the literature traditional immediate implant with immediate loading has high failure rate due to destructive horizontal forces, accordingly It was recommended for long time stress-free healing periods to achieve the osseointegration of dental implants.

But unfortunately this long time to restore the missing teeth is unsatisfactory to the patient due to high increase of patients' demand for perfect restoring missing teeth preservation of soft and hard tissues with better esthetic and functional results with decreasing the treatment plan time.

Rationale for conducting the research:

This study aimed to add a satellite implant device around the root form implant to enhance the primary implant stability for immediate loading followed by assessment of the final implant stability and final bone quantity and quality around the placed implant

DETAILED DESCRIPTION:
Research question:

Does the use of satellite implant technique for immediate loading will effectively reduce the treatment time without affection of the final implant stability and the final bone quality and quantity around the placed root form dental implant?

Statement of the problem:

Based on the literature traditional immediate implant with immediate loading has high failure rate due to destructive horizontal forces, accordingly It was recommended for long time stress-free healing periods to achieve the osseointegration of dental implants.

But unfortunately this long time to restore the missing teeth is unsatisfactory to the patient due to high increase of patients' demand for perfect restoring missing teeth preservation of soft and hard tissues with better esthetic and functional results with decreasing the treatment plan time.

Rationale for conducting the research:

This study aimed to add a satellite implant device around the root form implant to enhance the primary implant stability for immediate loading followed by assessment of the final implant stability and final bone quantity and quality around the placed implant

Review of literature:

A long time before there is increase of the patient demand for perfect restoring missing teeth with reducing the total time of treatment over all. So immediate loading implant was a very good solution especially in esthetic zone . However , it is not always applicable due to the difficult surrounding circumcenters Such like unfavorable type or quality of bone which makes immediate implant is impossible. Osseointegration of an implant, which is the main treatment goal, might best be understood to simply mean "undisturbed bone healing around the implant." Micro motion probably interferes with the development of an adequate early scaffold from the fibrin clot . Biomechanically, implants to be loaded immediately need to be stable and resistant to macro movement to ensure good osseointegration. Enhancement of implant stability can be achieved primarily by using a connecting bar as a stabilizer to provide a polygonal support to distribute forces and moments on single standing implants . This study aimed to add a satellite plate around the root form implant to enhance the primary implant stability for immediate loading followed by assessment of the final implant stability and final bone quantity and quality around the placed implant.

Objectives:

This study aimed to evaluate the final implant stability and bone condition after the use of satellite immediate implant with immediate loading in fresh extraction sockets.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking implant drive prosthesis after immediate extraction technique .
* Fresh extraction sockets with undestructed labial or palatal walls.
* Patients with non-restorable teeth due to untreatable caries or trauma.

Exclusion Criteria:

* General contraindications to implant surgery.
* Active infection or severe inflammation in the area intended for implant placement
* Teeth non restorable due to periodontal issues.
* Poor oral hygiene and motivation.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Patients participating in other studies, if the present protocol could not be properly followed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
final implant stability after satellite implant device removal. | 6 months
  OUT COME
  Calculate the final implant stability after plate removal.
  MEASURE DEVICE Osstell "resonance frequency analyzer"
  MEASURE UNIT ISQ

CONTACTS AND LOCATIONS:
Overall Officials: salah yassin, professor, Principal Investigator — • Professor of Oral and Maxillofacial Surgery, Faculty of Dentistry, Cairo University; Mohammed omaraa, lecturer, Study Director — • Lecturer in Oral and Maxillofacial Surgery- Cairo University.
Locations (1):
- Cairo university ,, Giza, Egypt